CLINICAL TRIAL: NCT06688448
Title: Comparative Efficacy and Durability of Next-Generation Biological Aortic Prostheses.
Brief Title: Valvular Assessment of New Generation Aortic Replacement Devices
Acronym: VANGUARD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto Dante Pazzanese de Cardiologia (Other)
Responsible Party: Principal Investigator, Tacianne Rolemberg Braga Delamain, Cardiologist assistant, Instituto Dante Pazzanese de Cardiologia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VANGUARD; Own resources (Other: Fundação Adib Jatene)
Record Dates: First submitted 2024-10-03; First posted 2024-11-14 (Actual); Last update posted 2025-01-13 (Actual); Status verified 2024-12

CONDITIONS: Aortic Regurgitation Disease; Aortic Valve Calcification; Bicuspid Aortic Valve Disease
Keywords: aortic valve surgery; Dafodil®; Inspires Resilia®; bioprosthetic valves; aortic valve replacement
MeSH Terms: conditions — Aortic Valve, Calcification of; Bicuspid Aortic Valve Disease

STUDY DESIGN:
Intervention Model Description: A prospective, open-label, single-center clinical study with randomization of 200 patients with indication of first-time or re-replacement aortic valve surgery to receive Dafodil® and Inspires Resilia® prostheses in the aortic position, conducted at a tertiary cardiology hospital of Brazilian Unified Health System (SUS)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Aortic Valve Replacement - Dafodil Prosthesis (Experimental): Patients indicated for surgical aortic valve replacement will be randomized to receive the Dafodil prosthesis.
  Interventions: Device: Dafodil prosthesis
- Aortic Valve Replacement - Inspires Resilia prosthesis (Active Comparator): Patients indicated for surgical aortic valve replacement will be randomized to receive Inspires Resilia prosthesis.
  Interventions: Device: Aortic Valve Replacement - Inspires Resilia prosthesis

INTERVENTIONS:
Device: Dafodil prosthesis — Surgical aortic valve replacement (SAVR) will be performed following standardized protocols to ensure consistency and optimize patient outcomes. Under general anesthesia, a median sternotomy will be conducted to access the aorta. Cardiopulmonary bypass (CPB) will be initiated, and the aorta will be cross-clamped to facilitate the safe removal of the existing prosthesis. After excising the deteriorated valve and removing any calcification, the new bioprosthetic valve will be implanted after randomized.
  Arms: Aortic Valve Replacement - Dafodil Prosthesis
Device: Aortic Valve Replacement - Inspires Resilia prosthesis — Surgical aortic valve replacement (SAVR) will be performed following standardized protocols to ensure consistency and optimize patient outcomes. Under general anesthesia, a median sternotomy will be conducted to access the aorta. Cardiopulmonary bypass (CPB) will be initiated, and the aorta will be cross-clamped to facilitate the safe removal of the existing prosthesis. After excising the deteriorated valve and removing any calcification, the new bioprosthetic valve will be implanted after randomized.
  Arms: Aortic Valve Replacement - Inspires Resilia prosthesis

SUMMARY:
The VANGUARD study is an open-label, prospective, randomized trial comparing the long-term outcomes of two advanced bioprosthetic aortic valves, Dafodil® and INSPIRIS Resilia®, in patients undergoing aortic valve replacement (AVR). This study aims to provide robust data on valve durability, safety, and hemodynamic performance, particularly in younger patients who may require multiple interventions over their lifetimes.

DETAILED DESCRIPTION:
This single-center, prospective open-label randomized clinical trial will enroll 200 patients indicated for aortic native valve or prosthetic valve replacement. Participants will be randomly assigned in a 1:1 ratio to receive the Dafodil® or INSPIRIS Resilia® prosthesis. The trial will be conducted at a leading tertiary cardiology hospital within the Brazilian Unified Health System (SUS). The study is sponsored by Instituto Dante Pazzanese de Cardiologia and Fundação Adib Jatene, with device supply supported by Meril Life Sciences (Vapi, Gujarat, India) and Edwards Lifesciences (Irvine, CA, USA).

Screening and Recruitment Process Participants will be identified through in-hospital referrals and outpatient clinics. The screening process will involve a comprehensive review of medical histories, imaging studies (e.g., echocardiograms), and relevant laboratory tests. To ensure a representative sample and minimize selection bias, the study will actively recruit patients with diverse comorbidities and histories of prior surgical procedures.

Informed Consent Process The informed consent process will adhere to stringent ethical standards, ensuring that participants fully understand the purpose, procedures, potential risks, and benefits of the study. The trained study personnel will provide detailed explanations and answer any questions. Patients will be informed of their right to withdraw from the study at any time without impacting their standard of care. Consent will be documented according to institutional guidelines.

Randomization and Blinding Participants will be randomized in a 1:1 ratio using the RedCap system , a secure web-based platform specifically designed for clinical trials. The randomization sequence will be generated using permuted blocks of varying sizes to maintain allocation concealment and ensure a balanced distribution across treatment groups.

Although the study is open-label due to the inherent nature of the surgical procedures, several strategies will be implemented to minimize bias:

* Outcome Adjudication and Imaging Assessment: Assessors responsible for evaluating postoperative echocardiographic imaging results and adjudicators of clinical outcomes will remain blinded to treatment allocation, thereby reducing the risk of observer bias.
* Centralized Data Monitoring: An independent team, blinded to treatment assignments, will conduct centralized data monitoring during audits and interim analyses, further safeguarding the study's integrity.
* Objective Outcome Measures: The study will prioritize objective measures, such as hemodynamic parameters and imaging findings, to minimize the potential influence of subjective bias.

Interventions Surgical Procedure: Surgical aortic valve replacement (SAVR) will be performed following standardized protocols to ensure consistency and optimize patient outcomes. Under general anesthesia, a median sternotomy will be conducted to access the aorta. Cardiopulmonary bypass (CPB) will be initiated, and the aorta will be cross-clamped to facilitate the safe removal of the existing prosthesis. After excising the deteriorated valve and removing any calcification, the new bioprosthetic valve-either Dafodil® or INSPIRIS Resilia®-will be implanted. Transesophageal echocardiography (TEE) will be utilized to assess valve function prior to weaning the patient off CPB. The procedure will conclude with the closure of the sternum and the patients transfer to the intensive care unit (ICU) for postoperative monitoring.

Postoperative Care: All patients will receive standardized postoperative care, encompassing anticoagulation management, pain control, and vigilant monitoring for potential complications. Follow-up assessments will include routine imaging and clinical evaluations to monitor recovery and verify the proper function of the implanted prosthesis. These evaluations will be scheduled at predetermined intervals to ensure timely detection and management of any issues that may arise.

Follow-up Schedule Participants will undergo follow-up evaluations at 30 days, 3 months, and annually for up to 10 years post-surgery. Each visit will encompass comprehensive data collection, including medical history updates, current medications, laboratory test results, electrocardiograms (ECGs), and echocardiograms. This structured follow-up schedule is designed to monitor patient recovery, assess the functionality of the implanted prosthesis, and promptly identify any emerging complications.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18 to 65 years.
* Eligible for surgical replacement of native valve or re-replacement of a prosthetic valve with a bioprosthetic valve in the aortic position.

Exclusion Criteria:

* Indicated for mechanical prosthetic valve replacement.
* Require surgical intervention in another heart valve or transcatheter valve therapy.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-12-01 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2036-12-01 (Estimated)

PRIMARY OUTCOMES:
Rate of bioprosthetic valve deterioration | 12 months
  Participants will be randomized equally to receive either the Dafodil® or INSPIRIS Resilia® valve. The primary outcome is Bioprosthetic valve deterioration, using the standardized definitions and will be assessed using survival analysis.

SECONDARY OUTCOMES:
Postoperative complications | 30 days
  Evaluate postoperative complications including hospitalization time, arrhythmias, bleeding, and surgical complications.
Quality of life | 10 years
  Quality of life will be assessed by The Kansas City Cardiomyopathy Questionnaire-12 (KCCQ-12). It is a simple, feasible, and sensitive questionnaire developed for assessing the health status composed of 4 domains: (1) physical limitation (items 1a, 1b, 1c), (2) symptom, frequency (items 2, 3, 4, 5), quality-of-life (items 6, 7), and social limitation (items 8a, 8b, 8c), [5] which are averaged to generate the Overall Summary score. Scores range from 0 to 100, with higher scores indicating fewer symptoms or limitations and better quality of life. To support its interpretation, cross-sectional scores of 0-24 indicate very poor to poor health status, 25-49 poor to fair, 50-74 fair to good, and 75-100 good to excellent health status. Changes of 5, 10, and ≥20 points indicate small but clinically important, moderate to large, and large to very large changes in patients' health status.
Treatment cost-effectiveness | 10 years
  Treatment cost-effectiveness will be assessed from the healthcare system perspective, focusing on time to valve deterioration and the need for subsequent procedures.

CONTACTS AND LOCATIONS:
Locations (1):
- Instituto Dante Pazzanese de Cardiologia, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No
IPD (Individual Patient Data) may not be shared due to concerns about patient confidentiality and data protection. Sharing such sensitive information could expose personal details and potentially violate privacy regulations. Additionally, there may be concerns about the misuse of data or its impact on the individuals privacy. Ensuring secure and ethical handling of IPD is crucial to protect patient rights and maintain trust.

REFERENCES:
- See also: Lasting durable bioprosthetic valves: Truth or fiction — https://doi.org/10.1016/j.xjon.2021.12.006
- See also: dized deﬁnitions of structural deterioration and valve failure in assessing long-term durability of transcatheter and surgical aortic bioprosthetic valves: a consensus statement from the European Association of Percutaneous Cardiovascular Interventions ( — https://pubmed.ncbi.nlm.nih.gov/28874031/
- See also: Prosthetic heart valves: selection of the optimal prosthesis and long-term management — https://pubmed.ncbi.nlm.nih.gov/19237674/
- See also: Update of the Brazilian Guidelines for Valvular Heart Disease - 2020 — https://pubmed.ncbi.nlm.nih.gov/33111877/
- See also: 2020 ACC/AHA Guideline for the Management of Patients With Valvular Heart Disease: Executive Summary: A Report of the American College of Cardiology/American Heart Association Joint Committee on Clinical Practice Guidelines — https://pubmed.ncbi.nlm.nih.gov/33342587/
- See also: 2021 ESC/EACTS Guidelines for the management of valvular heart disease: Developed by the Task Force for the management of valvular heart disease of the European Society of Cardiology (ESC) and the European Association for Cardio-Thoracic Surgery (EACTS) — https://pubmed.ncbi.nlm.nih.gov/35636831/